CLINICAL TRIAL: NCT02823977
Title: A Randomized, Double-blind Study of Ketamine / Dexmedetomidine vs. Placebo / Dexmedetomidine as Adjunctive Therapies for Severe Alcohol Withdrawal
Brief Title: Ketamine vs. Placebo as Adjunctive Therapies for Severe Alcohol Withdrawal
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding not obtained
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-1303
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Alcohol Withdrawal
Keywords: ketamine; dexmedetomidine; alcohol
MeSH Terms: interventions — Ketamine; Dexmedetomidine; Saline Solution; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine / Dexmedetomidine (Experimental): Ketamine 0.25 mg/kg bolus followed by 0.5 mg/kg per hour AND Dexmedetomidine by continuous infusion at a fixed rate of 0.6 µg/kg per hour, both administered for up to 72 hours
  Interventions: Drug: Ketamine; Drug: Dexmedetomidine
- Placebo / Dexmedetomidine (Placebo Comparator): Normal saline, as a 500 mL infusion bag, to represent placebo AND Dexmedetomidine by continuous infusion at a fixed rate of 0.6 µg/kg per hour, both administered for up to 72 hours
  Interventions: Drug: Dexmedetomidine; Drug: Normal saline

INTERVENTIONS:
Drug: Ketamine — Blinded study drug administered to experimental arm
  Other Names: Ketalar
  Arms: Ketamine / Dexmedetomidine
Drug: Dexmedetomidine — Open-label study drug administered to both arms
  Other Names: Precedex
Drug: Normal saline — Blinded comparator administered to control arm
  Other Names: 0.9% NaCl in water
  Arms: Placebo / Dexmedetomidine

SUMMARY:
This study is designed to evaluate the addition of ketamine to dexmedetomidine as adjunctive therapies of severe alcohol withdrawal in medical ICU patients. Specifically, this study will assess whether the combination of ketamine and dexmedetomidine reduces the doses of conventional agents used for alcohol withdrawal while maintaining patient comfort and safety and will explore if the combination alters the expression of catecholamines in the serum over time.

DETAILED DESCRIPTION:
The combination of ketamine and dexmedetomidine for alcohol withdrawal is pharmacologically rationale and may provide additive benzodiazepine-sparing effects. All subjects will receive benzodiazepine therapy as standard of care.

The objectives of this randomized, double-blind pilot study of 20 subjects with severe alcohol withdrawal are to a) determine if adding ketamine 0.5 mg/kg per hour to dexmedetomidine 0.6 µg/kg per hour (both agents administered for up to 72 hours) as adjunctive therapies to a symptom-triggered benzodiazepine protocol reduces the dose requirements of conventional sedatives while maintaining patient comfort and safety; and to b) explore whether epinephrine, a marker of autonomic activity, is expressed differently when ketamine is added to dexmedetomidine as adjunctive therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Severe alcohol withdrawal defined by a CIWA score ≥ 15 and the need for at least 16 mg of lorazepam equivalents over a four-hour period. All benzodiazepine and barbiturate doses, whether oral or intravenous, will contribute to the cumulative amount using the following conversion: 1 mg lorazepam = 2 mg midazolam = 7.5 mg clorazepate = 15 mg phenobarbital.
2. Patients receiving standard therapy for severe alcohol withdrawal according to the UCH-specific, symptom-triggered alcohol withdrawal protocol in the ICU (or admission to the ICU is anticipated). Lorazepam is the preferred benzodiazepine agent for patients requiring ICU admission due to alcohol withdrawal.
3. Informed consent within 36 hours of qualifying for the study.

Exclusion Criteria:

1. Patients < 18 years of age or > 85 years of age.
2. Patients receiving benzodiazepine therapy for purposes other than alcohol withdrawal (e.g. sedation, seizure control other than alcohol withdrawal).
3. Patients with alcohol withdrawal not requiring ICU admission.
4. Patients receiving epidural administration of medication(s).
5. Comatose patients by metabolic or neurologic affectation.
6. Patients with active myocardial ischemia or second- or third-degree heart block.
7. Patients with Child-Pugh score of C.
8. Moribund state with planned withdrawal of life support.
9. Patient pending transfer to another facility.
10. Patients with known or suspected severe adverse reactions to dexmedetomidine (or clonidine) or ketamine.
11. Pregnant females or females suspected of being pregnant.
12. Prisoners or active parolees.
13. Previous study participation.
14. Patients already receiving ketamine for alcohol withdrawal. Patients receiving dexmedetomidine will be excluded if the infusion exceeds 1 µg/kg per hour for more than two hours or any rate for a cumulative duration of 12 hours.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative Lorazepam Dose Over the First 12 Hours of Alcohol Withdrawal | 12 hours
  As part of routine care, the bedside nurse will record the administration of all sedative agents. The hourly, daily and cumulative doses of agents will be determined by the sum of as needed doses, scheduled intermittent doses, and hourly infusion rates. All conventional therapies will be guided by the institution-specific, symptom-triggered alcohol withdrawal protocol to maintain CIWA scores ≤ 7. Intravenous lorazepam is the preferred benzodiazepine for management of alcohol withdrawal in the medical ICU. Phenobarbital and propofol are infrequently used and they are not included in the protocol. All benzodiazepine and barbiturate doses, whether oral or intravenous, will be converted to lorazepam equivalents using the following conversion: 1 mg lorazepam = 2 mg midazolam = 7.5 mg clorazepate = 15 mg phenobarbital.
Cumulative Lorazepam Dose Over the First 24 Hours of Alcohol Withdrawal | 24 hours
  As part of routine care, the bedside nurse will record the administration of all sedative agents. The hourly, daily and cumulative doses of agents will be determined by the sum of as needed doses, scheduled intermittent doses, and hourly infusion rates. All conventional therapies will be guided by the institution-specific, symptom-triggered alcohol withdrawal protocol to maintain CIWA scores ≤ 7. Intravenous lorazepam is the preferred benzodiazepine for management of alcohol withdrawal in the medical ICU. Phenobarbital and propofol are infrequently used and they are not included in the protocol. All benzodiazepine and barbiturate doses, whether oral or intravenous, will be converted to lorazepam equivalents using the following conversion: 1 mg lorazepam = 2 mg midazolam = 7.5 mg clorazepate = 15 mg phenobarbital.
Cumulative Lorazepam Dose Over the 72 Hours of Alcohol Withdrawal | 72 hours
  As part of routine care, the bedside nurse will record the administration of all sedative agents. The hourly, daily and cumulative doses of agents will be determined by the sum of as needed doses, scheduled intermittent doses, and hourly infusion rates. All conventional therapies will be guided by the institution-specific, symptom-triggered alcohol withdrawal protocol to maintain CIWA scores ≤ 7. Intravenous lorazepam is the preferred benzodiazepine for management of alcohol withdrawal in the medical ICU. Phenobarbital and propofol are infrequently used and they are not included in the protocol. All benzodiazepine and barbiturate doses, whether oral or intravenous, will be converted to lorazepam equivalents using the following conversion: 1 mg lorazepam = 2 mg midazolam = 7.5 mg clorazepate = 15 mg phenobarbital.

SECONDARY OUTCOMES:
Change in 12-Hour Lorazepam Requirement Pre- and Post-Treatment | 12 hours before treatment, 12 hours after treatment on first day of starting study drug
  As part of routine care, the bedside nurse will record the administration of all sedative agents. The hourly, daily and cumulative doses of agents will be determined by the sum of as needed doses, scheduled intermittent doses, and hourly infusion rates. All conventional therapies will be guided by the institution-specific, symptom-triggered alcohol withdrawal protocol to maintain CIWA scores ≤ 7. Intravenous lorazepam is the preferred benzodiazepine for management of alcohol withdrawal in the medical ICU. Phenobarbital and propofol are infrequently used and they are not included in the protocol. All benzodiazepine and barbiturate doses, whether oral or intravenous, will be converted to lorazepam equivalents using the following conversion: 1 mg lorazepam = 2 mg midazolam = 7.5 mg clorazepate = 15 mg phenobarbital.
Change in 24-Hour Lorazepam Requirement Pre- and Post-Treatment | 24 hours before treatment, 24 hours after treatment on first day of starting study drug
  As part of routine care, the bedside nurse will record the administration of all sedative agents. The hourly, daily and cumulative doses of agents will be determined by the sum of as needed doses, scheduled intermittent doses, and hourly infusion rates. All conventional therapies will be guided by the institution-specific, symptom-triggered alcohol withdrawal protocol to maintain CIWA scores ≤ 7. Intravenous lorazepam is the preferred benzodiazepine for management of alcohol withdrawal in the medical ICU. Phenobarbital and propofol are infrequently used and they are not included in the protocol. All benzodiazepine and barbiturate doses, whether oral or intravenous, will be converted to lorazepam equivalents using the following conversion: 1 mg lorazepam = 2 mg midazolam = 7.5 mg clorazepate = 15 mg phenobarbital.
The Degree of Alcohol Withdrawal Assessed by Clinical Institute Withdrawal Assessment (CIWA) Scores | 72 hours
  CIWA scores will be assessed hourly by the bedside nurse. The proportion of CIWA scores ≥ 15 (severe withdrawal symptoms), 8 - 14 (moderate withdrawal symptoms), and ≤ 7 (minimal withdrawal symptoms) will be determined.
The Occurrence of Adverse Events: hypotension, hypertension, bradycardia, tachycardia | 72 hours
  Blood pressure and heart rate will be assessed hourly by the bedside nurse. Hypotension will be defined as a systolic blood pressure ≤ 90 mmHg or a decrease of systolic blood pressure of 40 mmHg, hypertension will be defined as a systolic blood pressure ≥ 180 mmHg or an increase of systolic blood pressure of 40 mmHg, bradycardia will be defined as a heart rate ≤ 55 beats/minute or a decrease of 20 beats/minutes, and tachycardia will be defined as a heart rate ≥ 120 beats/minute or an increase of 20 beats/minutes. Highest and lowest daily measurements of each will also be collected.
Plasma Epinephrine Concentrations Across Groups Over Time | 96 hours
  Plasma epinephrine concentrations will be assessed prior to study drug and at times 24, 48, 72 and 96 hours after initiating study drug

CONTACTS AND LOCATIONS:
Overall Officials: Robert MacLaren, PharmD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be presented and published in a peer reviewed journal. Individual data will not be shared.